CLINICAL TRIAL: NCT01142739
Title: A Descriptive Study of Lymphocytic Phosphorylation of ERK1/2 in Patients With Parkinson's Disease With Dyskinesias and in Controls
Brief Title: Phosphorylation of ERK1/2 in Patients With Parkinson's Disease
Acronym: BIODYS (1)
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2009/20
Record Dates: First submitted 2010-06-01; First posted 2010-06-11 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease patient: levodopa-treated parkinson's disease (PD) patients
  Interventions: Other: Clinical variables
- Non Parkinson's disease controls: Non Parkinson's disease controls
  Interventions: Other: Clinical variables

INTERVENTIONS:
Other: Clinical variables — Demography, disease duration, treatment duration, current treatment, daily intake of levodopa, Disease stage (Hoehn and Yahr, HY), motor score (UPDRS III) and dyskinesia severity (UPDRS IV). Biological variables.
  Groups: Parkinson's Disease patient
Other: Clinical variables — Demography, Biological variables.
  Groups: Non Parkinson's disease controls
Other: Clinical variables — Eye movement recordings : non-invasive infra-red camera oculometry (EyeBrain) before and after (only parkinson's disease group) levodopa(10 to 15 minute/recording)

SUMMARY:
Levodopa-induced dyskinesia severely limits the use of levodopa in Parkinson's disease and constitutes a debilitating complication of dopaminergic treatment in late stage. Among several neurobiological mechanisms identified so far, the investigators have established in experimental models the key role of D1 receptor hypersensitivity and a"Ras-ERK" signalling pathway. As the very same dopamine receptor machinery and the Ras-ERK pathway are present in blood lymphocytes, the investigators wish to test the hypothesis that the level of ERK phosphorylation in lymphocytes is a biomarker of levodopa-induced dyskinesia in Parkinson's Disease.

The study will be performed in dyskinetic levodopa-treated patients and non-Parkinson's Disease controls. Blood sampling "off" and "on" levodopa treatment (1 hour post-dose), as well as clinical data collection will be done during a scheduled pre-op work-up (deep brain stimulation). Subsequently, suspended lymphocytes from blood samples will be immunolabelled using an anti-pERK antibody and mean fluorescence intensity and percent of labelled lymphocytes will be assessed by flow cytometry. Additionally, plasma and urine samples will be collected "on" et "off" for dosage of dopamine. The motor effect of levodopa will be assessed through UPRSIII rating scale and eye movement (saccades) speed by non-invasive oculometric recordings.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive eligible PD in- and outpatients selected at the university hospital of Bordeaux.
* Non-demented patients (DSM IV) who are able to give their informed consent and who are affiliated to the social security.
* Controls: Subjects without known neurological disorder, non-demented, able to give their informed consent and affiliated to the social security.

Exclusion Criteria:

* Patients: Atypical or secondary parkinson disease.
* Previous or current cancer or malignant haemopathy.
* Known auto-immune disease.
* Anti-neoplastic or immuno-modulator treatment (particularly corticosteroids). Immuno-deficient subjects.
* Acute viral infection (within 2 weeks after resolving). Statin drug intake. Demented subject (DSMIV).
* Controls: Same criteria as above plus any neurological disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible PD in- and outpatients selected at the university hospital of bordeaux and subjects without known neurological disorder in a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
ERK phosphorylation | Day 1
  Distribution of variables and difference in the state of ERK phosphorylation in two contrasted groups : the dyskinetic levodopa-treated PD group and control group.

SECONDARY OUTCOMES:
plasma and urinary dopamine in "on" and "off" state | Day 1
measure derivatives of morphine | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie DAMON-PERRIERE, Dr., Principal Investigator — University Hospital, Bordeaux; Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux Hôpital Haut Lévêque, Pessac, France